CLINICAL TRIAL: NCT03793647
Title: Electrical Muscle Stimulation in Severely Deconditioned Congestive Heart Failure Patients- a Prospective, Randomized, Controlled Trial
Brief Title: Electrical Muscle Stimulation in Congestive Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Olten (Other)
Responsible Party: Principal Investigator, Nisha Arenja, Principle Investigator, Kantonsspital Olten
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-00273
Record Dates: First submitted 2018-10-05; First posted 2019-01-04 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Congestive Heart Failure; Electric Muscle Stimulation; Severe Decondition; Elderly Person; Exercise Capacity; Activities of Daily Living
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled study
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Intensity EMS (Active Comparator): Conventional Stimulation
  Interventions: Device: Electrical muscle devise
- High Intensity EMS (Experimental): Russian Stimulation
  Interventions: Device: Electrical muscle devise
- Placebo (Placebo Comparator): no Stimulation, supported by phone contact
  Interventions: Device: Electrical muscle devise

INTERVENTIONS:
Device: Electrical muscle devise — evaluate two types of EMS stimulation of legs

SUMMARY:
This trial is to evaluate two types of electrical muscle Stimulation (EMS) stimulation (low intensity "conventional stimulation" vs. high intensity "Russian" stimulation) of legs in comparison with a control group without EMS in a cohort of elderly patients with severe deconditioning after CHF decompensation.

DETAILED DESCRIPTION:
BACKGROUND:

Congestive heart failure (CHF) is increasingly prevalent worldwide and is associated with significant morbidity and mortality. Poor exercise capacity is well known as a risk factor for poor prognosis. The deconditioning is mainly associated with a decrease in leg muscle mass and loss of leg strength as well as loss of muscle endurance. This affects especially elderly patients. To improve this condition in CHF electrical muscle stimulation (EMS) is a suitable method of training, which hardly affects the heart. However, most EMS existing stimulation protocols are uncomfortable and not user-friendly, especially for elderly patients. The Russian space medicine has many years' experience in specific EMS stimulation protocols, which are well tolerated by cosmonauts for hours even during working activities. Therefore, a research project has been established between the Russian Academy of Sciences (Laboratory for Biomedical Problems) and the ARTORG Research Center for Biomedical Engineering to study the effects of new developed EMS procedures in elderly persons.

Aims:

The aim of trial is to evaluate two types of EMS stimulation (low intensity "conventional stimulation" vs. high intensity "Russian" stimulation) of legs in comparison with a control group without EMS in a cohort of elderly patients with severe deconditioning after CHF decompensation.

METHOTOLOGY:

This prospective, randomized controlled study will use commercially available electronic stimulator devices (Medel GmbH, Hamburg, Germany) for EMS. For the "Russian" stimulation, an especial developed stimulator (Amplidin-EST No.5) will be used for frequency modulation of the stimulation impulse, which is supposed to make stimulation sensation more comfortable. Supervised EMS training will be performed 5 times per week (weekdays) during 30 minutes over a period of 6 weeks in elderly deconditioned CHF patients, starting at the Kantonsspital Olten during the hospitalisation and continued at home. We will include 20 patients in each group (20 in control group, 20 in low intensity "conventional group and 20 in high intensity "Russian" group). The control group was preformed to exclude an attention bias in the study results. The primary endpoint of the study is the difference in maximum oxygen uptake (peak VO2) and in 6 minutes walking distance between baseline and after 6-weeks EMS training in all groups (high intensity vs low intensity vs control). The follow-up period is planned for 2 years.

POTENTIAL SIGNIFICANCE:

Exercise capacity and quality of life in severely deconditioned patients with CHF is poor and life expectancy is low. While the possibilities to improve the poor condition and function of the heart by pharmaceutical therapies are limited, there is potential to improve the condition of the peripheral muscles by exercise training. However, a successful aerobic training is rarely feasible in these patients. Therefore, EMS training may prove to be ideal tool to improve leg muscle mass and function of elderly patients. Because, CHF patients do not tolerate most of the existing EMS stimulation protocols, we have developed a new EMS stimulation protocol. The application is virtually painless and therefore well tolerated over hours due to a sophisticated stimulation protocol. Therefore, we hope that, this especial for elderly CHF patients developed training protocol, may improve their daily activity as well as their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* hospitalized due to heart failure
* left ventricular ejection fraction ≤ 40%
* NYHA class II to IV
* willingness to complete the 6-week EMS training programme
* tolerability of the electrical stimulation
* provision of informed consent

Exclusion Criteria:

* severe neuromuscular or oncologic diseases with inability to perform exercise testing and EMS training
* inotropic intravenous agents used (≤10 days)
* implanted pacemaker/ICD
* unstable angina
* severe uncontrolled arrhythmias
* patients with severe pulmonary limitation (Tiffeneau ratio <70%, or vital capacity <70% of predicted value)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in 6 minutes walking distance after EMS training | 2 years
  The primary outcome of the study is the difference in 6 minutes walking distance (m) between baseline and after 6-weeks EMS training in all groups (high intensity vs low intensity vs control).

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Arenja, Principal Investigator — Kantonsspital Olten
Locations (1):
- Kantonsspital Olten, Olten, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deley G, Kervio G, Verges B, Hannequin A, Petitdant MF, Salmi-Belmihoub S, Grassi B, Casillas JM. Comparison of low-frequency electrical myostimulation and conventional aerobic exercise training in patients with chronic heart failure. Eur J Cardiovasc Prev Rehabil. 2005 Jun;12(3):226-33. doi: 10.1097/01.hjr.0000166455.23346.a5. PMID 15942420
- [Background] Dobsak P, Novakova M, Siegelova J, Fiser B, Vitovec J, Nagasaka M, Kohzuki M, Yambe T, Nitta S, Eicher JC, Wolf JE, Imachi K. Low-frequency electrical stimulation increases muscle strength and improves blood supply in patients with chronic heart failure. Circ J. 2006 Jan;70(1):75-82. doi: 10.1253/circj.70.75. PMID 16377928
- [Background] Harris S, LeMaitre JP, Mackenzie G, Fox KA, Denvir MA. A randomised study of home-based electrical stimulation of the legs and conventional bicycle exercise training for patients with chronic heart failure. Eur Heart J. 2003 May;24(9):871-8. doi: 10.1016/s0195-668x(02)00822-9. PMID 12727155
- [Background] Karavidas A, Arapi SM, Pyrgakis V, Adamopoulos S. Functional electrical stimulation of lower limbs in patients with chronic heart failure. Heart Fail Rev. 2010 Nov;15(6):563-79. doi: 10.1007/s10741-010-9171-9. PMID 20490656
- [Background] Karavidas A, Driva M, Parissis JT, Farmakis D, Mantzaraki V, Varounis C, Paraskevaidis I, Ikonomidis I, Pirgakis V, Anastasiou-Nana M, Filippatos G. Functional electrical stimulation of peripheral muscles improves endothelial function and clinical and emotional status in heart failure patients with preserved left ventricular ejection fraction. Am Heart J. 2013 Oct;166(4):760-7. doi: 10.1016/j.ahj.2013.06.021. Epub 2013 Aug 30. PMID 24093858
- [Background] Nuhr M, Crevenna R, Gohlsch B, Bittner C, Pleiner J, Wiesinger G, Fialka-Moser V, Quittan M, Pette D. Functional and biochemical properties of chronically stimulated human skeletal muscle. Eur J Appl Physiol. 2003 Apr;89(2):202-8. doi: 10.1007/s00421-003-0792-8. Epub 2003 Feb 28. PMID 12665986
- [Background] Quittan M, Sochor A, Wiesinger GF, Kollmitzer J, Sturm B, Pacher R, Mayr W. Strength improvement of knee extensor muscles in patients with chronic heart failure by neuromuscular electrical stimulation. Artif Organs. 1999 May;23(5):432-5. doi: 10.1046/j.1525-1594.1999.06372.x. PMID 10378936
- [Background] Sbruzzi G, Ribeiro RA, Schaan BD, Signori LU, Silva AM, Irigoyen MC, Plentz RD. Functional electrical stimulation in the treatment of patients with chronic heart failure: a meta-analysis of randomized controlled trials. Eur J Cardiovasc Prev Rehabil. 2010 Jun;17(3):254-60. doi: 10.1097/HJR.0b013e328339b5a2. PMID 20560163
- [Background] Smart NA, Dieberg G, Giallauria F. Functional electrical stimulation for chronic heart failure: a meta-analysis. Int J Cardiol. 2013 Jul 15;167(1):80-6. doi: 10.1016/j.ijcard.2011.12.019. Epub 2012 Jan 10. PMID 22236510
- [Background] Vaquero AF, Chicharro JL, Gil L, Ruiz MP, Sanchez V, Lucia A, Urrea S, Gomez MA. Effects of muscle electrical stimulation on peak VO2 in cardiac transplant patients. Int J Sports Med. 1998 Jul;19(5):317-22. doi: 10.1055/s-2007-971924. PMID 9721054